CLINICAL TRIAL: NCT01033786
Title: Recovery After Robotic Urogynecological Surgery: Hospital Stay and Perioperative Complications of Patients Who Did Not Complete Questionnaires
Brief Title: Robotic Urogynecological Surgery: Hospital Stay and Perioperative Complications
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: 29966
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Urogynecology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess length of hospital stay and perioperative complications of patients undergoing daVinci Robot-assisted sacrocolpopexy, during a one-year time period, who did not complete a questionnaire on post-operative recovery.

ELIGIBILITY:
Inclusion Criteria:

* The first 21 women who underwent DaVinci-assisted robotic sacrocolpopexy and who did not complete postoperative QA questionnaires from 09/01/2007 through 09/01/2008.

Exclusion Criteria:

* Any women not meeting inclusion criteria.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who underwent DaVinci-assisted laparscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2009-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To assess length of hospital stay and perioperative complications of patients undergoing daVinci Robot-assisted sacrocolpopexy, during a one-year time period, who did not complete a questionnaire on post-operative recovery. | 09/01/07 - 09/01/08

CONTACTS AND LOCATIONS:
Overall Officials: Gunhilde Buchsbaum, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States